CLINICAL TRIAL: NCT02765022
Title: Clip Closure of Mucosal Defects After Endoscopic Mucosal Resection of Large Colorectal Lesions as Prophylaxis of Delayed Haemorrhage.
Brief Title: Clip Closure of Mucosal Defects After Endoscopic Mucosal Resection.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMSALBE
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2018-08

CONDITIONS: Endoscopic Resection; Clip; Haemorrhage; Non-pedunculated Lesions
MeSH Terms: conditions — Hemorrhage | interventions — Surgical Instruments

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Clip (Experimental): Clip closure of mucosal defects after endoscopic mucosal resection.
  Interventions: Device: Clip closure
- No clip (Active Comparator): No clip closure of mucosal defects after endoscopic mucosal resection. Observation.
  Interventions: Procedure: No clip closure

INTERVENTIONS:
Device: Clip closure — Complete clip closure of secondary lesions after the endoscopic mucosal resection
  Arms: Clip
Procedure: No clip closure — Observation: no clip closure of secondary lesions after the endoscopic mucosal resection
  Arms: No clip

SUMMARY:
An simple-blind, randomized study, to evaluate the efficacy and safety of complete closure with clips of mucosal defects after endoscopic mucosal resection (EMR) of large non-pedunculated colorectal lesions (≥ 2 cm) as prophylaxis of delayed bleeding.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Clinical indication of endoscopic mucosal resection for large-sized (≥ 2cm) non-pedunculated colorectal lesions.
* Medium-high risk of delayed bleeding (DB risk score ≥ 4)
* Informed consent.

Exclusion Criteria:

* Patients with colorectal non-pedunculated lesions without endoscopic mucosal resection indication.
* Lesions resected by endoscopic submucosal resection.
* Incomplete resections.
* Resections with suspected deep submucosal invasion.
* Mucosal defects treated with clips for known or suspected damage to the muscle layer.
* Lesions with low risk of delayed bleeding (DB risk score ≤3).
* Patients with any other medical, geographic or social condition, deemed by the Investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interfere with the interpretation of the results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Delayed hemorrhage | 15 days post-EMR

CONTACTS AND LOCATIONS:
Locations (1):
- Eduardo Albeniz Arbizu, Pamplona, Navarre, Spain

REFERENCES:
- [Derived] Albeniz E, Alvarez MA, Espinos JC, Nogales O, Guarner C, Alonso P, Rodriguez-Tellez M, Herreros de Tejada A, Santiago J, Bustamante-Balen M, Rodriguez Sanchez J, Ramos-Zabala F, Valdivielso E, Martinez-Alcala F, Fraile M, Elosua A, Guerra Veloz MF, Ibanez Beroiz B, Capdevila F, Enguita-German M. Clip Closure After Resection of Large Colorectal Lesions With Substantial Risk of Bleeding. Gastroenterology. 2019 Nov;157(5):1213-1221.e4. doi: 10.1053/j.gastro.2019.07.037. Epub 2019 Jul 27. PMID 31362007
- See also: Related Info — http://navarrabiomed.es